CLINICAL TRIAL: NCT06829719
Title: Personalization of Maintenance Immunosuppression Based on TTV Viral Load to Prevent Long-term Complications in Renal Transplantation
Brief Title: TTV-based mAnagement Of Long-term ImmunosuppreSsion in Kidney Transplantation
Acronym: TAOIST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Collaborators: BioMérieux (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 69HCL23_0834
Record Dates: First submitted 2025-02-03; First posted 2025-02-17 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-02

CONDITIONS: Infection; Cancer; Rejection; Kidney Transplantation
Keywords: TTV; Biomarker; immunosuppression; precision medicine; kidney transplantation
MeSH Terms: conditions — Infections; Neoplasms; Rejection, Psychology

STUDY DESIGN:
Intervention Model Description: Prospective, interventional, multicentric, open-label, parallel group, superiority randomized controlled trial.
  Kidney transplant recipients from the 4 enrollment centers will be randomly assigned with a 1:1 allocation into experimental and control groups between 12- and 48-months post-transplantation, and prospectively followed for 36 months for the occurrence of a complication due to inadequate (over or under) immunosuppression.
Who Masked: Investigator
Masking Description: TTV DNAemia will be measured every 3 months for all patients but the results will not be communicated to the physicians for patients from the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TTV-guided immunosuppression (Experimental): The adaptation of the dose of maintenance immunosuppressive drugs will be based on TTV DNAemia measured on site in the plasma of patients every 3 months (at distance of an infection or a vaccination). The physicians will be free to change the dose of calcineurin inhibitors (CNI) and/or the mycophenolate mofetil (MMF) to maintain TTV DNAemia between 3.8 and 5.1 log10 cp/mL as long as the trough levels remain between 3-12 ng/mL for tacrolimus (50-250 ng/mL for cyclosporin) and the daily dose of MMF is comprise between 250 and 1500 mg bid for Cellcept (180 and 900 mg for Myfortic).
  Interventions: Biological: TTV DNAemia; Other: EQ-5D-5L questionnaire; Biological: Biological tests
- Standard Immunosuppression (Other): TTV DNAemia will also be measured every 3 months but the results will not be communicated to the physicians. Instead, the adaptation of the dose of maintenance immunosuppressive drugs will be performed according to the current standard of care: i) the dose of the CNI will be adapted to maintain the trough levels, monitored in the circulation every 3 month, between 5-10 ng/mL for tacrolimus (75-150 ng/mL for cyclosporin) and ii) the dose of MMF will be adjusted to maintain the AUC, measured every year, between 30-60 h.mg/L.
  Interventions: Biological: TTV DNAemia; Other: EQ-5D-5L questionnaire; Biological: Biological tests

INTERVENTIONS:
Biological: TTV DNAemia — Every 3 months, one sample added at the same time (7mL) of a routine laboratory analysis for TTV DNAemia
Other: EQ-5D-5L questionnaire — Completed every 6 months and each time a complication of interest occurs
Biological: Biological tests — Biological tests as routine care procedure (creatinine, CNI pre-dose trough level) will be performed every 6 months

SUMMARY:
Long-term outcomes in kidney transplantation remain a significant challenge, as complications such as donor-specific antibodies (DSA), antibody-mediated rejection, infections, and cancer increasingly threaten graft and patient survival over time. The development of non-invasive biomarkers to guide the management of therapeutic immunosuppression beyond the first year post-transplantation is therefore a crucial unmet need.

Torque Teno Virus (TTV), a non-pathogenic virus with a high prevalence worldwide, has emerged as a promising biomarker in this context. Its replication inversely reflects immune control by T cells, correlating with the depth of therapeutic immunosuppression. Additionally, its slow replication kinetics make TTV DNAemia a useful marker for evaluating patient adherence to immunosuppressive treatments.

The TAOIST study tests whether longitudinal monitoring of TTV DNAemia every three months, starting from the second year after transplantation, can guide the personalization of immunosuppressive therapy. The primary endpoint is the time to the first occurrence of complications linked to inadequate immunosuppression, including dnDSA, biopsy-proven rejection, infection, cancer, or graft loss. Secondary objectives include evaluating the acceptability of TTV DNAemia among healthcare professionals and assessing its cost-effectiveness compared to standard care. An ancillary objective examines the link between TTV DNAemia and the immunosuppressant possession ratio (IPR) to explore its potential as a marker of treatment adherence.

ELIGIBILITY:
Inclusion Criteria:

* Adult ≥ 18 years-old
* Recipient of a kidney allograft (third graft at most)
* 12 to 48 months post-transplantation
* Stable graft function (defined as: delta creatininemia over the previous 6 months < 20% and proteinuria < 30mg/mmol)
* On maintenance immunosuppression, which includes CNI (cyclosporin or tacrolimus) and MMF (Cellcept or Myfortic) with or without corticosteroids
* Detectable TTV DNAemia at enrollment
* No circulating DSA in solid phase assay
* Undetectable BKV DNAemia at enrollment
* Written informed consent

Exclusion Criteria:

* Recipient of an HLA identical graft
* Mutiple organ transplantation or functional transplant other than kidney
* Maintenance immunosuppression that includes a mTOR inhibitor, belatacept or imurel
* Presence of histological sign of active rejection (i+t > 2 and g+cpt > 2) on graft biopsy performed within 3 months before enrollment
* Uncontrolled infection at inclusion
* Infection requiring hospitalization or vaccination within 3 months before inclusion
* Pregnant, unwillingness to practice adequate contraception or patient with a pregnancy plan during 3 years of study
* Person not affiliated to a social security scheme or beneficiary of a similar scheme
* Person subject to a legal protection measure (guardianship, curatorship) or deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-04-23 (Actual); Primary Completion 2028-05-01 (Estimated); Study Completion 2031-02-02 (Estimated)

PRIMARY OUTCOMES:
Compare the time from inclusion to first complication of inadequate immunosuppression between the experimental group, whose treatment is tailored on quarterly TTV viral load results, and the control group. | through study completion, an average of 6 years
  Time from inclusion to occurrence of the first complication of inadequate immunosuppression: development of dnDSA, biopsy-proven rejection, infection, cancer, graft loss. Patients lost to follow-up or died without an event before will be right censored at this date.

SECONDARY OUTCOMES:
Proportion of patients with at least one complication of inadequate immunosuppression between the experimental and control groups at 36 months | through study completion, an average of 6 years
  Percentage of patients with at least one complication of inadequate immunosuppression during the 36 months of follow-up.
Compare the rate of complications of inadequate immunosuppression between patients in the experimental and control groups. | through study completion, an average of 6 years
  Number of complications of inadequate immunosuppression/patient/month of follow-up
Describe the nature and timing of various complications of inadequate immunosuppression in the experimental and control groups. | through study completion, an average of 6 years
  Percentage of patients (at 36 months) and time to first complication for each of the complications of interest: development of dnDSA, biopsy-proven rejection, infection, cancer, graft loss.
Compare the proportion of patients with adequate immunosuppressive therapy between the experimental and control groups. | through study completion, an average of 6 years
  Percentage of patients with TTV viral load between 3.8 and 5.1 log cp/ml at the majority (>6/12) of quarterly routine controls.
Compare the proportion of quarterly systematic checks of TTV DNAemia in the target between patients in the experimental and control groups. | Every 3 months
  Percentage of quarterly routine TTV viral load tests between 3.8 and 5.1 log cp/ml.
Model the impact of variations in dose and residual rates (pre-dose trough levels or AUC) of the various immunosuppressive drugs on TTV viral load. | every 3 months
  Joint analysis of the evolution of dose variations, residual immunosuppression rates of immunosuppressive drugs and TTV viral load.
Evaluate how nephrologists and biologists feel about using the new test in clinical practice. | 6th year
  Questionnaires specific to each sub-populations (nephrologists and biologists) using open-ended questions and Likert scale-coded responses.
Assess the cost-effectiveness of the intervention compared to standard care at 36 months from the French Health care System perspective | through study completion, an average of 6 years
  Cost-effectiveness ratio (ICER) is defined as the difference in cost between the intervention and the standard care, divided by the difference in their effect (QALY).

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Service de Néphrologie-Transplantation-Dialyse I Hôpital Pellegrin I - CHU Bordeaux, Bordeaux (France)
  - Service de transplantation, néphrologie et immunologie clinique Hospices Civils de Lyon, Hôpital Edouard Herriot, Lyon
  - Service de Néphrologie, Dialyse et Transplantation Rénale Nouvel Hôpital Civil, Strasbourg (france)
  - Département de Néphrologie et Transplantation d'Organes Hôpital Rangueil - CHU de Toulouse, Toulouse (France)